CLINICAL TRIAL: NCT06366139
Title: Comparison of the Efficacy of Trigeminal Ganglion Radiofrequency Thermocoagulation and Ultrasound-guided Maxillary-mandibular Pulsed Radiofrequency in the Treatment of Trigeminal Neuralgia
Brief Title: Trigeminal Ganglion RFT vs Maxillary/Mandibular PRF in the Treatment of Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Supervisor Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Trigeminal RFT vs max/mand PRF
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Trigeminal Neuralgia; Headache Disorders
Keywords: Pulsed Radiofrequency Treatment; Radiofrequency Ablation; Maxillary Nerve; Mandibular Nerve
MeSH Terms: conditions — Trigeminal Neuralgia; Headache Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiofrequency thermocoagulation group (Active Comparator): Trigeminal ganglion radiofrequency thermocoagulation for trigeminal neuralgia
  Interventions: Procedure: Radiofrequency thermocoagulation of the trigeminal ganglion
- pulsed radiofrequency group (Active Comparator): Maxillary mandibular nerve pulsed radiofrequency for trigeminal neuralgia
  Interventions: Procedure: Maxillary/Mandibular nerve pulsed radiofrequency

INTERVENTIONS:
Procedure: Radiofrequency thermocoagulation of the trigeminal ganglion — The patient is placed in the supine position and the foramen ovale is identified medial to the coronoid process of the mandible by giving the head a submental oblique position under fluoroscopic guidance. A 20-gauge, 5 mm active type, and 100 mm radiofrequency cannula is inserted 2 cm lateral to the commissura labialis and advanced towards the foramen. After entering the foramen ovale with a lateral fluoroscopic image, the radiofrequency cannula is connected to the radiofrequency generator and sensory and motor stimulations are performed to confirm the target maxillary and mandibular nerves. The radiofrequency lesion is applied at 60°C, 65°C and 70°C for 60-seconds periods. The patient is observed for side effects for 1 hour after the procedure.
  Arms: radiofrequency thermocoagulation group
Procedure: Maxillary/Mandibular nerve pulsed radiofrequency — The patient is placed in the lateral decubitus position with the affected side up. A 5-12 MHz linear ultrasound probe is placed in the infrazygomatic area above the maxilla at a 45° inclination in both the frontal and horizontal planes. The probe position allows visualization of the pterygopalatine fossa, which is limited to the maxilla anteriorly and the greater wing of the sphenoid posteriorly. Real-time ultrasound guidance allows direct localization of the internal maxillary artery and identification of the needle tip. The radiofrequency cannula was connected to the radiofrequency generator and PRF was applied at 42°C for 240 seconds after confirming the localization of the maxillary and mandibular nerve by obtaining appropriate responses to sensory and motor stimulation.
  Arms: pulsed radiofrequency group

SUMMARY:
Trigeminal ganglion (TG) radiofrequency thermocoagulation (RFT) and ultrasound (US)-guided maxillary or mandibular (max/mand) pulsed radiofrequency (PRF) are two interventional procedures for the treatment of trigeminal neuralgia (TN). The aim of this study was to compare the efficacy and safety of these two procedures. For this evaluation, the numeric rating scale (NRS) was used to assess pain relief and the Medication Quantification Scale III (MQS III) was used to assess the effectiveness of the interventions on medication consumption. The rates of adverse events related to the interventions were also compared.

DETAILED DESCRIPTION:
Trigeminal neuralgia (TN) is a very severe, unilateral, short, lightning-like pain that starts and ends suddenly and is limited to the areas related to the branches of the trigeminal nerve. The pain can be triggered by stimuli such as washing face, shaving, smoking, talking and/or brushing teeth (trigger factors) and usually occurs spontaneously.

Treatment of TN is complex despite the use of multiple medications and may be resistant. Interventional procedures are an option in cases that do not respond to medical treatments or if there are side effects. Interventional procedures include trigeminal ganglion RFT and maxillary-mandibular (max/mand) nerve PRF. PRF delivers short bursts of high-voltage electrical current to the target nerve, creating a non-thermal effect that modulates the transmission of pain signals. RFT delivers a continuous current that heats the target tissue, causing coagulation necrosis on nerves.

Although trigeminal ganglion RFT is a frequently performed method in the treatment of idiopathic TN, there is limited literature data on ultrasonography (US)-guided max/mand nerve PRF.

The primary aim of this study was to compare the efficacy of trigeminal ganglion RFT and max/mand nerve PRF for TN. Secondary aims were to determine the effects of interventions on drug consumption and interventional safety based on adverse events. A total of at least 44 patients, 22 patients in each group, will be enrolled for comparison. NRS, and MQS III scores before treatments, 1 month, and 6 months after treatments will be compared both within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic TN according to the international headache society
* Pain for at least 6 months and numeric rating scale (NRS) score greater than 6 despite medical treatment (despite the maximum tolerated dose of carbamazepine, gabapentinoid or tramadol)

Exclusion Criteria:

* Vascular compression of the trigeminal nerve by MRI and MRI angiography and the presence of secondary causes such as multiple sclerosis
* Dental or temporomandibular joint pathologies
* Previous interventional procedures or surgery for TN
* Coagulopathy or use of antiaggregants and anticoagulants
* Cardiac pacemaker
* Renal-hepatic insufficiency
* Diagnosis of psychiatric illness
* Malignancy and
* Injection site or systemic infection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-02-04 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) | Change from baseline to 1st and 6th month after treatment
  NRS is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain)

SECONDARY OUTCOMES:
The Medication Quantification Scale III (MQS III) | Change from baseline 6th month after treatment
  The MQS III is a validated tool in medical research that quantifies medication regimens by assigning a numerical value to each medication based on its class, dosage, and associated risks. This scale aids clinicians and researchers in tracking changes in pain levels throughout a treatment course or study, providing an objective measure of medication consumption and its potential negative impact.

CONTACTS AND LOCATIONS:
Overall Officials: Gevher Rabia Genc Perdecioğlu, Study Chair — Diskapi TRH
Locations (1):
- Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)